CLINICAL TRIAL: NCT05096117
Title: Human Laboratory Study of ASP8062 for Alcohol Use Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLAB-003
Record Dates: First submitted 2021-10-19; First posted 2021-10-27 (Actual); Results first posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Alcohol Use Disorder; Alcohol Drinking; Alcohol Use Disorder (AUD)
MeSH Terms: conditions — Alcoholism; Alcohol Drinking | interventions — ASP8062

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ASP8062 (25 mg once daily) (Experimental)
  Interventions: Drug: ASP8062
- Matching Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP8062 — ASP8062 is a novel compound with positive allosteric modulator (PAM) activity on the γ-aminobutyric acid type B (GABAB) receptor, 25 mg, 1 x per day for 6 weeks
  Arms: ASP8062 (25 mg once daily)
Drug: Placebo — 1 x per day for 6 weeks
  Arms: Matching Placebo

SUMMARY:
The primary objective of this study is to evaluate the effects of ASP8062, 25 mg once a day and matched placebo, on alcohol cue-elicited alcohol craving during a human laboratory paradigm after 2 weeks of daily dosing among subjects with moderate to severe alcohol use disorder (AUD) as confirmed by the Diagnostic and Statistical Manual of Mental Disorders - Fifth Edition (DSM-5™). Secondary objectives include evaluation of ASP8062, 25 mg once a day, and matched placebo on reduction of alcohol consumption, alcohol craving, cigarette smoking (among smokers), mood, sleep, alcohol use negative consequences, study retention, and safety and tolerability throughout the last 4 weeks of the treatment phase of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 21 years of age.
2. Meet the DSM-5 criteria for AUD of at least moderate severity.
3. Be seeking treatment for AUD and desire a reduction or cessation of drinking.
4. Be able to verbalize an understanding of the consent form, able to provide written informed consent, verbalize willingness to complete study procedures, able to understand written and oral instructions in English and able to complete the questionnaires required by the protocol.
5. Agree (if the subject is female and of child bearing potential) to use at least one of the following methods of birth control to at least 30 days post the last dose of study drug, unless she is surgically sterile, partner is surgically sterile or she is postmenopausal (one year):

   1. oral contraceptives,
   2. contraceptive sponge,
   3. patch,
   4. double barrier (diaphragm/spermicidal or condom/spermicidal),
   5. intrauterine contraceptive system,
   6. etonogestrel implant,
   7. medroxyprogesterone acetate contraceptive injection,
   8. true abstinence: when this is in line with the preferred and usual lifestyle of the participant,
   9. and/or hormonal vaginal contraceptive ring.
6. Agree (if female) to not donate ova for at least 30 days following the last ASP8062 administration.
7. Agree (if male) to use acceptable methods of contraception if the male participant's partner could become pregnant from the time of the first administration of the study drug until 90 days following the final administration of the study drug. One of the following acceptable methods of contraception must be utilized:

   1. surgical sterilization (vasectomy);
   2. the participant's female partner uses oral contraceptives (combination estrogen/progesterone pills), injectable progesterone or sub dermal implants (commenced at least 14 days prior to study drug administration to the male participant)
   3. the participant's female partner uses a medically prescribed topically applied transdermal contraceptive patch (commenced at least 14 days prior to study drug administration to the male participant);
   4. the participant's female partner has undergone tubal ligation (female sterilization) or is postmenopausal (one year);
   5. the participant's female partner has undergone placement of an intrauterine device or intrauterine system; and,
   6. true abstinence: when this is in line with the preferred and usual lifestyle of the participant.
8. Agree (if male) to refrain from sperm donation from the randomization visit to at least 90 days after the last dose of study drug.
9. Be able to take oral medication and be willing to adhere to the medication regimen.
10. Complete all assessments required at screening and baseline.
11. Have a place to live in the 2 weeks prior to randomization and not be at risk that s/he will lose his/her housing in the next 2 months.

    Not anticipate any significant problems with transportation arrangements or available time to travel to the study site over the next 2 months.
12. Not have any unresolved legal problems that could jeopardize continuation or completion of the study.
13. Provide contact information of someone, such as a family member, spouse, or significant other, who may be able to contact the subject in case of a missed clinic appointment.
14. Have a BAC by breathalyzer equal to 0.000 when s/he signed the informed consent document.
15. If taking a medication for depression or anxiety, must have been taking a stable dose in the 2-months prior to randomization and plan to continue during the study. This includes drugs such as the following:

    1. Selective serotonin reuptake inhibitors (SSRIs)
    2. Dual uptake inhibitors
    3. Serotonin-norepinephrine reuptake inhibitors (SNRIs)
    4. Tricyclic antidepressants
16. Be someone who in the opinion of the investigator would be expected to complete the study protocol.
17. Agree to the schedule of visits, verbally acknowledge that s/he will be able to attend each scheduled visit, participate in phone visits and that s/he does not have any already scheduled events or a job that may substantially interfere with study participation.
18. Be willing to use a smartphone's video capability to record daily oral ingestion of tablets for the entire 6-week treatment period (subject's own smartphone or one provided by AiCure).
19. Have sitting (3 to 5 minutes) vital signs at the screening visit within the following limits:

    1. Systolic blood pressure 90 to 140 mmHg
    2. Diastolic blood pressure of 50 to 90 mmHg
    3. Heart rate of 40 to 90 beats per minute

Exclusion Criteria:

1. Current (past 12 months) substance use disorder of at least moderate severity (4 or more criteria) for any psychoactive substance other than alcohol and nicotine, including sedatives and hypnotics, or cocaine use disorder of any severity as defined by DSM-5 criteria.
2. Be mandated by the court to obtain treatment for alcohol-dependence, or has probation or parole requirements that might interfere with study participation.
3. Be anyone who in the opinion of the investigator could not be safely withdrawn from alcohol without medical detoxification.
4. Have any of the following, based on DSM-5 criteria as assessed using theMINI:

   1. Current or lifetime diagnosis of psychotic disorders,
   2. Current bipolar disorder,
   3. Current major depressive episode,
   4. Current (past 3 months) eating disorder (anorexia or bulimia), or
   5. Within past year diagnosis of panic disorder with or without agoraphobia.

Contact site for additional exclusion criteria.

-

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2023-03-22 (Actual); Study Completion 2023-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raye Litten, Ph.D., Study Director — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (3):
- United States (3):
  - University of California Los Angeles, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - Brown University, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
Data and supporting information will be shared with the general research community upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available approximately 6/25/2025 for an indefinite time period
Access Criteria: Data users will be encouraged to complete a Data Use Agreement and obtain authorization for data use by the NIAAA Data Access Committee.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ASP8062 (25 mg Once Daily) | Matching Placebo
Started | 30 | 30
Completed | 28 | 26
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ASP8062 (25 mg Once Daily) | Matching Placebo | Total
Number analyzed (Participants) | 28 | 26 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (9.8) | 45.4 (10.0) | 43.8 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 20
  Male | 16 | 18 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 18 | 20 | 38
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 28 | 26 | 54
Drinks per week [Mean (Standard Deviation); unit: Standard drinks of alcohol/week] | 53.5 (22.1) | 52.3 (20.1) | 52.9 (21.0)

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Craving
Description: Strength of alcohol craving Visual Analogue Scale (VAS) score; min=0, max=20; higher scores = more craving (worse outcome)
Time Frame: Week 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | ASP8062 (25 mg Once Daily) | Matching Placebo
Number analyzed (Participants) | 28 | 26
score on a scale | 6.44 (1.09) | 6.26 (1.13)
Statistical Analysis 1: Comparison: ASP8062 (25 mg Once Daily) vs Matching Placebo; Test type: Superiority; p = 0.784, ANCOVA; Least Square Mean Difference = .178

2. Secondary Outcome: Number of Subjects With no Heavy Drinking Days
Description: Number of subjects that have no heavy drinking days during weeks 3 to 6 of the treatment phase. A "heavy drinking day" is 4 or more drinks per drinking day for women and 5 or more drinks per drinking day for men.
Time Frame: Weeks 3 to 6 of the treatment phase
Measure: Count of Participants; unit: Participants
Arm/Group | ASP8062 (25 mg Once Daily) | Matching Placebo
Number analyzed (Participants) | 28 | 26
Participants | 2 | 1

3. Secondary Outcome: Number of Subjects Abstinent From Alcohol
Description: Number of subjects that have not drank alcohol during Weeks 3 to 6 of the treatment phase.
Time Frame: Weeks 3 to 6 of the treatment phase
Measure: Count of Participants; unit: Participants
Arm/Group | ASP8062 (25 mg Once Daily) | Matching Placebo
Number analyzed (Participants) | 28 | 26
Participants | 0 | 1

4. Secondary Outcome: WHO 1-level Decrease in Alcohol Consumption
Description: The number of subjects experiencing at least a 1-level decrease in World Health Organization (WHO) levels of alcohol consumption from the level at baseline (the period including the 28 days before screening) to the level during Weeks 3 to 6 of the treatment phase.
  The WHO levels of average alcohol consumption per day are as follows:
  Males Females Low Risk 1 to 40g 1 to 20g Medium Risk 41 to 60g 21 to 40g High Risk 61 to 100g 41 to 60g Very High Risk 101+g 61+g where 14g = 1 SDU (WHO-2000). In computing the WHO alcohol consumption level, average drinks per day were used, computed as the sum of all drinks in the 28 day period divided by the number of days with non-missing drinking data in that period. Abstinent subjects were included in a separate "Abstinent" category.
Time Frame: Weeks 3 to 6 of the treatment phase
Measure: Count of Participants; unit: Participants
Arm/Group | ASP8062 (25 mg Once Daily) | Matching Placebo
Number analyzed (Participants) | 28 | 26
Participants | 19 | 18

5. Secondary Outcome: WHO 2-level Decrease in Alcohol Consumption
Description: The number of subjects experiencing at least a 2-level decrease in World Health Organization (WHO) levels of alcohol consumption from the level at baseline (the period including the 28 days before screening) to the level during Weeks 3 to 6 of the treatment phase.
  The WHO levels of average alcohol consumption per day are as follows:
  Males Females Low Risk 1 to 40g 1 to 20g Medium Risk 41 to 60g 21 to 40g High Risk 61 to 100g 41 to 60g Very High Risk 101+g 61+g where 14g = 1 SDU (WHO-2000). In computing the WHO alcohol consumption level, average drinks per day were used, computed as the sum of all drinks in the 28 day period divided by the number of days with non-missing drinking data in that period. Abstinent subjects were included in a separate "Abstinent" category.
Time Frame: Weeks 3 to 6 of the treatment phase.
Measure: Count of Participants; unit: Participants
Arm/Group | ASP8062 (25 mg Once Daily) | Matching Placebo
Number analyzed (Participants) | 28 | 26
Participants | 8 | 11

6. Secondary Outcome: Percentage of Days Abstinent
Description: The percentage of days abstinent from drinking alcohol
Time Frame: Weeks 3 to 6 of the treatment phase
Measure: Least Squares Mean (Standard Error); unit: percentage of days abstinent
Arm/Group | ASP8062 (25 mg Once Daily) | Matching Placebo
Number analyzed (Participants) | 28 | 26
percentage of days abstinent | 29.9 (5.4) | 39.3 (5.6)

7. Secondary Outcome: Percentage of Heavy Drinking Days
Description: Percentage of heavy drinking days where a heavy drinking day is 4 or more drinks on a day for women or 5 or more drinks on a day for men.
Time Frame: Weeks 3 to 6 of the treatment phase
Measure: Least Squares Mean (Standard Error); unit: percentage of heavy drinking days
Arm/Group | ASP8062 (25 mg Once Daily) | Matching Placebo
Number analyzed (Participants) | 28 | 26
percentage of heavy drinking days | 42.4 (6.1) | 35.9 (6.3)

8. Secondary Outcome: Drinks Per Week
Description: The number of drinks consumed per week
Time Frame: Weeks 3 to 6 of the treatment phase
Measure: Least Squares Mean (Standard Error); unit: standard drinks of alcohol/week
Arm/Group | ASP8062 (25 mg Once Daily) | Matching Placebo
Number analyzed (Participants) | 28 | 26
standard drinks of alcohol/week | 28.2 (4.0) | 23.7 (4.1)

9. Secondary Outcome: Drinks Per Drinking Day
Description: The number of drinks consumed on days where participants drank
Time Frame: Weeks 3 to 6 of the treatment phase
Measure: Least Squares Mean (Standard Error); unit: standard drinks of alcohol/drinking day
Arm/Group | ASP8062 (25 mg Once Daily) | Matching Placebo
Number analyzed (Participants) | 28 | 26
standard drinks of alcohol/drinking day | 5.7 (0.5) | 5.5 (0.5)

10. Secondary Outcome: Penn Alcohol Craving Scale (PACS)
Description: The amount of craving; higher numbers indicate more craving. There are 5 items each on a 0 to 6 scale. Items are summed to get to the total craving, resulting in scores having a min=0 and max=30.
Time Frame: Weeks 3 to 6 during the treatment phase, averaged
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | ASP8062 (25 mg Once Daily) | Matching Placebo
Number analyzed (Participants) | 28 | 26
score on a scale | 13.5 (0.9) | 13.0 (1.0)

11. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI)
Description: A measure of sleep quality; the PSQI includes a scoring key for calculating a patient's seven subscores, each of which can range from 0 to 3. The subscores are tallied, yielding a "global" score that can range from 0 to 21. A global score of 5 or more indicates poor sleep quality; the higher the score, the worse the quality.
Time Frame: Weeks 4 & 6 of the treatment phase, averaged
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | ASP8062 (25 mg Once Daily) | Matching Placebo
Number analyzed (Participants) | 28 | 26
score on a scale | 5.7 (0.4) | 6.1 (0.4)

12. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Alcohol Related Negative Consequences
Description: A measure of alcohol-related negative consequences. There are 7 items scored on a 1 to 7 scale (a higher score indicative greater frequency of negative consequences). The items are summed and converted to a T-score to create a total score. The T-scores range from 0 to 100 (the population mean = 50 and standard deviation = 10). Higher T-scores are indicative of more negative consequences (worse outcome).
Time Frame: Week 6 of the treatment phase
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | ASP8062 (25 mg Once Daily) | Matching Placebo
Number analyzed (Participants) | 28 | 26
T-score | 50.2 (1.0) | 47.8 (1.1)

13. Secondary Outcome: Profile of Mood States (POMS) Total Disturbance
Description: A measure of total mood disturbance. Total mood disturbance is the sum of depression, anger, fatigue, confusion, and tension subscales subtracting the vigor subscale items. The range of possible scores is from -32 to 200 with higher scores indicating greater mood disturbance.
Time Frame: Weeks 4 & 6 of the treatment phase, averaged
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | ASP8062 (25 mg Once Daily) | Matching Placebo
Number analyzed (Participants) | 28 | 26
score on a scale | 5.0 (3.6) | 0.5 (3.8)

14. Secondary Outcome: Cigarettes Smoked Per Day (Among Smokers)
Description: The number of cigarettes smoked per day, computed among individuals who smoked at baseline
Time Frame: Weeks 3 to 6 of the treatment phase
Measure: Least Squares Mean (Standard Error); unit: cigarettes smoked per day
Arm/Group | ASP8062 (25 mg Once Daily) | Matching Placebo
Number analyzed (Participants) | 28 | 26
cigarettes smoked per day | 10.3 (1.2) | 10.7 (2.0)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | ASP8062 (25 mg Once Daily) | Matching Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 24/30 | 22/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASP8062 (25 mg Once Daily) (N=30) | Matching Placebo (N=30)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bundle branch block right (Cardiac disorders) | 0 (0) | 1 (1)
Conduction disorder (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 2 (2)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (5) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (3) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Influenza like illness (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 1 (1)
Blood albumin increased (Investigations) | 0 (0) | 1 (1)
Blood alkaline phosphatase decreased (Investigations) | 0 (0) | 2 (2)
Blood bicarbonate decreased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Blood cholesterol increased (Investigations) | 4 (4) | 2 (2)
Blood creatinine decreased (Investigations) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 0 (0)
Blood urine present (Investigations) | 1 (1) | 0 (0)
Electrocardiogram T wave abnormal (Investigations) | 0 (0) | 1 (1)
Glucose urine present (Investigations) | 1 (1) | 1 (1)
Protein urine (Investigations) | 4 (4) | 2 (2)
Red blood cell count decreased (Investigations) | 1 (1) | 1 (1)
Red cell distribution width increased (Investigations) | 1 (1) | 0 (0)
Triglyceride analyses (Investigations) | 1 (1) | 0 (0)
Urine ketone body present (Investigations) | 1 (1) | 2 (2)
Urine leukocyte esterase positive (Investigations) | 2 (2) | 2 (2)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 4 (5) | 2 (2)
Headache (Nervous system disorders) | 3 (5) | 4 (6)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 4 (4) | 2 (2)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (3)
Blunted affect (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (6)
Irritability (Psychiatric disorders) | 1 (2) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (1) | 1 (1)
Stress (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (2) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 10 (17) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-08-12): https://cdn.clinicaltrials.gov/large-docs/17/NCT05096117/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-13): https://cdn.clinicaltrials.gov/large-docs/17/NCT05096117/SAP_001.pdf
  • Informed Consent Form (2022-03-24): https://cdn.clinicaltrials.gov/large-docs/17/NCT05096117/ICF_002.pdf